CLINICAL TRIAL: NCT07182825
Title: Evaluation of the Effects of Multifidus Lift Exercise on Endurance, Pain, and Disability in University Students With Low Back Pain
Brief Title: Effects of Multifidus Lift Exercise on Endurance, Pain, and Disability in University Students With Low Back Pain
Acronym: LBP-MULEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Guler (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Mehmet Akif Guler, PhD, Lecturer, Selcuk University
Organization: Selcuk University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUTUBITAK996; 1919B012413996 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Non Specific Chronic Low Back Pain; Healthy Vollunteer
Keywords: Nonspecific Low Back Pain; Multifidus Muscle; Multifidus Lift Exercise; Bird-Dog Exercise (Modified); Spinal Stabilization Exercise; Endurance; Pain; Disability; Oswestry Disability Index (ODI); Visual Analog Scale (VAS); Biering-Sørensen Test; University Students; Young Adults; Healthy Controls
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Intervention Model Description: Two parallel groups will be studied: (1) university students aged 18-25 years with nonspecific chronic low back pain, and (2) healthy controls without low back pain. Both groups will receive the same 6-week supervised modified Multifidus Lift Exercise protocol. Group allocation is based on participants' clinical status; no randomization will be performed.
Masking Description: No masking will be implemented. Both participants and investigators are aware of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSCLBP Students - Modified Multifidus Lift Exercise (Experimental): University students aged 18-25 years with nonspecific chronic low back pain. Participants will perform the supervised modified Multifidus Lift Exercise protocol, twice weekly for 6 weeks. Each session includes warm-up, exercise progression (8-15 repetitions depending on week), and cool-down. Outcomes: lumbar extensor endurance (primary), pain intensity (VAS), and functional disability (ODI).
  Interventions: Behavioral: Modified Multifidus Lift Exercise (MLE)
- Healthy Students - Modified Multifidus Lift Exercise (Experimental): Healthy university students aged 18-25 years without low back pain in the past 3 months. Participants will perform the same supervised modified Multifidus Lift Exercise protocol, twice weekly for 6 weeks, with identical warm-up, exercise progression, and cool-down. Outcome: lumbar extensor endurance (Biering-Sørensen Test).
  Interventions: Behavioral: Modified Multifidus Lift Exercise (MLE)

INTERVENTIONS:
Behavioral: Modified Multifidus Lift Exercise (MLE) — A supervised stabilization exercise protocol designed to selectively activate the lumbar multifidus muscle. In the quadruped position, the contralateral knee is maintained approximately 10 cm above the ground while the participant performs controlled trunk stabilization. Sessions are conducted twice weekly for 6 weeks, each including warm-up (5 minutes brisk walk, mobilization, hamstring stretch), the modified Multifidus Lift Exercise with progressive repetitions (weeks 1-2: 8-10, weeks 3-4: 10-12, weeks 5-6: 12-15), and cool-down (static stretches). All sessions are supervised to ensure correct form, breathing control, and safety.
  Other Names: Modified Bird-Dog Exercise; Multifidus Lift

SUMMARY:
Nonspecific low back pain is a common musculoskeletal problem that also affects many young adults, including university students. It can negatively impact academic performance, daily life, and overall well-being. Research shows that stabilization exercises targeting the lumbar multifidus muscle play an important role in rehabilitation, but it is unclear whether modified versions of these exercises may provide additional benefits.

This study will investigate a simple modification of the traditional "bird-dog" exercise, called the "Multifidus Lift Exercise." In this version, participants maintain the contralateral knee about 10 cm above the ground while in a four-point kneeling position. This adjustment is expected to increase multifidus activation and improve back endurance.

University students aged 18-25 with nonspecific low back pain will participate in a 6-week supervised program, performing the exercise twice weekly. A healthy control group without low back pain will also be included. The main outcome will be back extensor muscle endurance (Biering-Sørensen Test). In participants with back pain, pain intensity (Visual Analog Scale) and functional disability (Oswestry Disability Index) will also be measured.

The study aims to determine whether this low-cost, practical, and time-efficient exercise can improve muscle endurance, reduce pain, and decrease disability in young adults with low back pain. Results may provide evidence for an effective and accessible preventive and therapeutic approach in student populations.

DETAILED DESCRIPTION:
Background and Rationale. Nonspecific low back pain (NSLBP) is highly prevalent in young adults and is associated with decreased academic performance, daily activity limitations, and reduced well-being. Stabilization exercises targeting segmental control-particularly the lumbar multifidus-are widely supported in rehabilitation literature. Conventional four-point kneeling ("bird-dog") activates multifidus and erector spinae; however, whether targeted modifications can yield greater multifidus activation remains insufficiently studied. This study evaluates a simple, low-cost modification termed the "Multifidus Lift Exercise" (MLE): in quadruped, the contralateral knee is maintained ~10 cm off the ground to bias multifidus recruitment. We hypothesize that MLE will improve lumbar extensor endurance and, in participants with NSLBP, reduce pain and disability.

Objectives and Research Questions. Primary objective: determine the effect of a 6-week supervised MLE program (2 sessions/week) on lumbar extensor endurance (Biering-Sørensen test). Secondary objectives (NSLBP group): assess changes in pain (10-cm VAS) and functional disability (Oswestry Disability Index, Turkish validated version). Key research questions test whether MLE increases endurance and reduces pain/disability in NSLBP, and whether endurance differs between NSLBP and healthy students.

Design and Setting. Single-center, interventional, non-randomized, parallel-group, pre-post design conducted at the Physiotherapy & Rehabilitation Exercise Hall, Selçuk University (Konya, Türkiye). Two cohorts will be observed under the same intervention protocol: (1) university students (18-25 y) with NSLBP and (2) healthy controls without recent low back pain. Allocation is based on current status (no randomization). Masking is not feasible (exercise behavior). Primary purpose: treatment/rehabilitation.

Intervention (Exercise Protocol). All participants receive an initial brief training on isolated multifidus activation and motor control principles. Each supervised session includes standardized warm-up (5 min brisk walk; mobilization; hamstring stretch), the MLE performed slowly and with breath control, and cool-down (static stretches). Repetition progression: weeks 1-2: 8-10 reps; weeks 3-4: 10-12; weeks 5-6: 12-15, emphasizing form and endurance. A 3-week pilot (2 sessions/week) mirrors the 6-week protocol in compressed form (wk1→8-10; wk2→10-12; wk3→12-15) to estimate effect size for main-study sample size planning.

Outcomes and Assessments. Primary outcome is Biering-Sørensen endurance time (seconds) in both groups. Secondary outcomes in NSLBP include VAS pain and ODI (%). Measurements occur at baseline and post-intervention. Adverse symptoms prompting immediate pause (e.g., dizziness, undue fatigue) are recorded session-wise.

See "Outcome Measures" and "Time Frame" modules for exact definitions and schedules.

Participants and Eligibility. Target population: Selçuk University students aged 18-25. Two cohorts (NSLBP vs healthy) are defined by clinical status and physician clearance for exercise. Inclusion/exclusion criteria address red flags, recent surgery or neurological deficits, pregnancy, regular analgesic use, high-load sports, and recent structured exercise that could confound endurance.

Complete criteria are provided in the "Eligibility" module.

Sample Size and Pilot-Informed Planning. The pilot (n≈20; 10 NSLBP/10 healthy) will provide effect size estimates (Cohen's d) to power the main study via G*Power. The anticipated main-study enrollment will be balanced across cohorts per power analysis.

Statistical Analysis (Summary). Analyses will use two-tailed α=0.05 with 95% CIs (IBM SPSS). Descriptives will summarize baseline characteristics. Normality will guide test selection. Between-group comparisons for endurance (NSLBP vs healthy) will use t-test or Mann-Whitney U. Within-group pre-post changes (endurance for both groups; VAS/ODI for NSLBP) will use paired t-tests or Wilcoxon signed-rank. Where appropriate, repeated-measures ANOVA (with Greenhouse-Geisser adjustment) will model time effects; ANCOVA may adjust for baseline imbalances. Exploratory Pearson/Spearman correlations will assess relationships among endurance, pain, and disability; multiple linear regression may evaluate predictors of disability change.

Safety and Monitoring. This is a low-risk, behavioral exercise intervention. Sessions are supervised by study staff; standardized stop rules (e.g., onset of dizziness, dyspnea, undue fatigue, new pain flare) are applied. A formal Data Monitoring Committee is not planned; safety is monitored by the investigative team at each session. Adverse events and withdrawals are documented.

Ethics and Oversight. Ethics approval was granted by the Selçuk University Faculty of Health Sciences Ethics Committee for Non-Interventional Clinical Investigations (Decision/Approval No: 2025/674; Meeting No: 05; Ref: 2025/05; Date: 30/04/2025). Participation is voluntary with written informed consent. Data are handled under the Declaration of Helsinki and applicable regulations (including Turkish KVKK). De-identified, aggregate results will be disseminated.

Data Handling and Dissemination. De-identified data will be analyzed and reported in aggregate. Individual participant data sharing is not planned. Findings will be prepared for peer-reviewed publication and scientific meetings, and may inform practical, community-oriented exercise programs for student populations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years

Currently enrolled as a university student at Selçuk University

Willing to participate voluntarily and sign informed consent form

Medically suitable for exercise participation

For NSCLBP group:

History of nonspecific chronic low back pain within the past 3 months

Physician confirmation of nonspecific low back pain

Oswestry Disability Index (ODI) ≥ 21% (moderate disability)

Visual Analog Scale (VAS) score ≥ 3.5

For Healthy control group:

No history of low back pain within the past 3 months

Physician confirmation of no contraindications for exercise

Exclusion Criteria:

* Presence of radicular pain or nerve root compression symptoms

History of spinal surgery

Neurological deficits within the past 3 months (e.g., muscle weakness, reflex loss, paresthesia)

Systemic infection or systemic disease affecting participation

Cardiovascular or pulmonary disease contraindicating exercise

Clinical "red flag" symptoms (e.g., saddle anesthesia, bowel/bladder incontinence, fever, known cancer)

Pregnancy

Regular use of analgesics, muscle relaxants, or anti-inflammatory medications

Participation in regular exercise programs in the past 3 months

Active involvement in sports directly affecting lumbar muscles (e.g., fitness, pilates, yoga, swimming)

Inability to comply with exercise sessions or study protocol

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Lumbar Extensor Muscle Endurance (Biering-Sørensen Test) | Baseline (pre-test) and after 6 weeks of intervention.
  Endurance of the lumbar extensor muscles will be assessed using the standardized Biering-Sørensen Test. Participants lie prone with the upper body unsupported beyond the table edge while the pelvis and lower limbs are stabilized. The duration (in seconds) that the participant can maintain the horizontal position without >10° deviation is recorded.

SECONDARY OUTCOMES:
Pain Intensity (Visual Analog Scale, VAS) | Baseline (pre-test) and after 6 weeks of intervention.
  Pain intensity will be measured using a 10-cm Visual Analog Scale, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Participants in the NSCLBP group will mark their pain level on the scale, and the distance (cm) from the "no pain" anchor will be recorded.
Functional Disability (Oswestry Disability Index, ODI) | Baseline (pre-test) and after 6 weeks of intervention.
  The Oswestry Disability Index (ODI) will be used to assess the impact of low back pain on daily living. It consists of 10 items scored 0-5, with higher scores indicating greater disability. The total score will be converted into a percentage. Only participants in the NSCLBP group will complete the ODI.

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision on IPD sharing will be made after study completion and in accordance with institutional and ethical guidelines

REFERENCES:
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Stevens VK, Vleeming A, Bouche KG, Mahieu NN, Vanderstraeten GG, Danneels LA. Electromyographic activity of trunk and hip muscles during stabilization exercises in four-point kneeling in healthy volunteers. Eur Spine J. 2007 May;16(5):711-8. doi: 10.1007/s00586-006-0181-1. Epub 2006 Aug 1. PMID 16896840
- [Background] Smeets R, Koke A, Lin CW, Ferreira M, Demoulin C. Measures of function in low back pain/disorders: Low Back Pain Rating Scale (LBPRS), Oswestry Disability Index (ODI), Progressive Isoinertial Lifting Evaluation (PILE), Quebec Back Pain Disability Scale (QBPDS), and Roland-Morris Disability Questionnaire (RDQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S158-73. doi: 10.1002/acr.20542. No abstract available. PMID 22588742
- [Background] Shafshak TS, Elnemr R. The Visual Analogue Scale Versus Numerical Rating Scale in Measuring Pain Severity and Predicting Disability in Low Back Pain. J Clin Rheumatol. 2021 Oct 1;27(7):282-285. doi: 10.1097/RHU.0000000000001320. PMID 31985722
- [Background] Sarafadeen R, Ganiyu SO, Ibrahim AA. Effects of spinal stabilization exercise with real-time ultrasound imaging biofeedback in individuals with chronic nonspecific low back pain: a pilot study. J Exerc Rehabil. 2020 Jun 30;16(3):293-299. doi: 10.12965/jer.2040380.190. eCollection 2020 Jun. PMID 32724788
- [Background] Pitcher MJ, Behm DG, Mackinnon SN. Neuromuscular fatigue during a modified biering-sorensen test in subjects with and without low back pain. J Sports Sci Med. 2007 Dec 1;6(4):549-59. eCollection 2007. PMID 24149491
- [Background] Pirouzi S, Emami F, Taghizadeh S, Ghanbari A. Is Abdominal Muscle Activity Different from Lumbar Muscle Activity during Four-Point Kneeling? Iran J Med Sci. 2013 Dec;38(4):327-33. PMID 24293787
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Demoulin C, Vanderthommen M, Duysens C, Crielaard JM. Spinal muscle evaluation using the Sorensen test: a critical appraisal of the literature. Joint Bone Spine. 2006 Jan;73(1):43-50. doi: 10.1016/j.jbspin.2004.08.002. PMID 16461206
- [Background] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- See also: Güler MA, Demirdel E, Albayrak İ, Nayman A. The Relationship between Core Stability, Pain and Disability in Persons with Chronic Non-Specific Low Back Pain. Selçuk Sağlık Dergisi. 2023;4(3):420-431. — https://dergipark.org.tr/en/pub/ssd/issue/82496/1363638#article_cite